CLINICAL TRIAL: NCT07339020
Title: Cyanoacrylate Versus Omentum for Enforcement of the Staple Line in Sleeve Operation
Brief Title: Cyanoacrylate Versus Omentum for Staple-Line Reinforcement in Sleeve Gastrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Eid Ali Ahmed Aziz, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ms-199-2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Bariatric surgery; Cyanoacrylate; Glubran; Laparoscopic sleeve gastrectomy; Omentopexy; Staple Line Reinforcement; Postoperative Hemorrhage; Surgical Leak
MeSH Terms: conditions — Obesity; Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: cyanoacrylate sealant (Glubran®) (Experimental): Group A: the reinforcement of staple line was done by cyanoacrylate sealant (Glubran®) from the angle of His till the lower end using its applicator through the right working port
  Interventions: Device: Glubran® 2 surgical glue (n-butyl-2-cyanoacrylate mixture) and its specific applicator.; Procedure: Staple Line Reinforcement during Laparoscopic Sleeve Gastrectomy
- Group B: Omentopexy (Active Comparator): Group B: the reinforcement was done by suturing the greater omentum to the staple line using PDS 2/0 round.
  Interventions: Biological: Autologous Greater Omentum; Procedure: Staple Line Reinforcement during Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Device: Glubran® 2 surgical glue (n-butyl-2-cyanoacrylate mixture) and its specific applicator. — A synthetic surgical adhesive applied to the staple line for reinforcement and hemostasis using its proprietary delivery applicator.
  Arms: Group A: cyanoacrylate sealant (Glubran®)
Biological: Autologous Greater Omentum — pedicled flap of the patient's own greater omentum sutured over the staple line for reinforcement using a PDS 2/0 round needle suture.
  Arms: Group B: Omentopexy
Procedure: Staple Line Reinforcement during Laparoscopic Sleeve Gastrectomy — Reinforcement of the gastric staple line during laparoscopic sleeve gastrectomy.

SUMMARY:
Study Title:

Comparing Surgical Glue (Cyanoacrylate) vs. Omentum Tissue to Strengthen Staple Lines in Weight-Loss Sleeve Surgery

What is the purpose of this study? This study will compare two ways to strengthen the staple line during weight-loss sleeve surgery. One way uses a medical glue called cyanoacrylate, and the other uses a piece of tissue from the abdomen called omentum. The goal is to see which method works better to lower the chance of bleeding, pain, or leaks after surgery.

Who can take part?

Adults ages 18-65 who:

* Have a body mass index (BMI) over 35, or over 30 if they also have health problems related to obesity.
* Are scheduled to have weight-loss sleeve surgery at Cairo University Hospital.

Participants cannot take part if they:

* Are younger than 18 or older than 65.
* Have had weight-loss surgery before.

What will happen in the study?

* Participants will be assigned by chance to one of two groups:

  1. Glue group: The staple line will be sealed with medical glue.
  2. Omentum group:The staple line will be covered and sewn with a piece of the body's own tissue.
* Everyone will have the same type of surgery and be cared for in the same way afterward.
* Participants will be monitored closely for one month after surgery to check for problems like bleeding, pain, or leaks.
* Follow-up visits will happen within one week after surgery and again at one month.

What are the possible risks? The risks are low and similar to those of regular weight-loss surgery. Some people may feel pain or anxiety after surgery. The study team will watch for any problems and treat them right away.

Why is this study being done? Weight-loss sleeve surgery is common, but sometimes the staple line can leak or bleed. Finding a better way to strengthen it may help people recover more safely and with less pain.

How long will the study last? The study will take about six months to complete, including surgery and follow-up.

Who is running the study? The study is being done by doctors in the General Surgery Department at Cairo University's Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Cases underwent LSG with age ≥18 years old and ≤65 years old and BMI ≥35 or ≥30 with comorbid disease related to obesity.
* Candidate for Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

* Cases underwent previous bariatric surgery.
* Multiple Extensive previous surgeries.
* Crohn's Disease.
* Elderly patients with extensive comorbidities
* Severe gastroesophageal reflux disease (GERD)
* Severe Bleeding disorders
* Psychiatric illness or cognitive impairment affecting consent or compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of Staple Line Complications After Sleeve Gastrectomy: Glubran vs. Omentum | From surgery up to 30 days postoperatively
  This measure compares two methods of staple line reinforcement during laparoscopic sleeve gastrectomy to see which works better at preventing complications within the first 30 days after surgery. The complications of interest are postoperative leakage (staple line leak), bleeding requiring intervention, and abdominal pain. Patients are randomly assigned to have their staple line reinforced either with medical glue (cyanoacrylate) or with the patient's own fatty tissue (omentum).

SECONDARY OUTCOMES:
Comparison of Operative Time Between Reinforcement Methods | Measured on the day of surgery.
  This measure compares the total surgical time (in hours) from skin incision to closure between the two study groups: cyanoacrylate glue reinforcement vs. omentum reinforcement.
Length of Hospital Stay After Sleeve Gastrectomy | From surgery until discharge, assessed up to 30 days postoperatively.
  This measure compares the number of days patients stay in the hospital after surgery between the two reinforcement groups, from the day of surgery until discharge.
Economic Cost of Reinforcement Materials | Assessed on the day of surgery
  This measure compares the direct cost of the reinforcement materials used in each group: cyanoacrylate glue versus omentum
Incidence of Delayed Staple Line Complications | From discharge up to 30 days postoperatively.
  This measure assesses whether any staple line complications (such as delayed leakage or bleeding) occur after discharge, within the first month post-surgery.
Rate of Hospital Readmission Within 30 Days | Within 30 days after discharge.
  This measure compares the proportion of patients in each group who are readmitted to the hospital within 30 days after discharge due to any surgery-related complication.
Rate of Reoperation Within 30 Days | Within 30 days postoperatively.
  This measure compares the proportion of patients in each group who require a second surgical intervention (reoperation) within 30 days after the initial surgery due to complications such as bleeding, leakage, or hematoma.

OTHER OUTCOMES:
Postoperative Pain Intensity Assessment | Daily from day of surgery up to 7 days postoperatively.
  This measure compares patient-reported pain levels (using a visual analog scale, VAS) (VAS, 0-10) during the first 7 days after surgery between the cyanoacrylate and omentum reinforcement groups.
Postoperative Nausea and Vomiting (PONV) Incidence | From end of surgery up to 48 hours postoperatively.
  This measure compares the incidence and severity of postoperative nausea and vomiting (PONV) in the first 48 hours after surgery between the two reinforcement groups.
Time to First Oral Intake | From end of surgery up to 48 hours.
  This measure compares the time (in hours) from end of surgery to first tolerated oral fluid intake (sips of water) between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Al-Manial Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No